CLINICAL TRIAL: NCT00292201
Title: Pilot Study of Statin Treatment in Patients With Stable Moderate to Severe Asthma
Brief Title: Statin Treatment in Patients With Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding to complete subject recruitment and testing
Sponsor: Queen's University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Ontario Lung Association (Other)
Responsible Party: Principal Investigator, Dr. Diane Lougheed, Professor, Department of Medicine, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 120973
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Asthma
Keywords: Asthma; Statin
MeSH Terms: conditions — Asthma | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Atorvastatin
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator): Placebo Pill
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — The treatment group will receive Atorvastatin 80 mg po once per day for 4 weeks. The placebo group will receive an identical placebo pill po once per day for 4 weeks.
  Other Names: Lipitor

SUMMARY:
Asthma is a chronic respiratory condition characterized by bronchial hyper-responsiveness secondary to abnormal inflammation of the lung. Steroids remain the most effective treatment for this condition. The lipid lowering agents statins have been found to have anti-inflammatory properties. This study is to test the hypothesize that statins will decrease bronchial hyperresponsiveness and inflammation, leading to improved symptoms in patients with asthma.

DETAILED DESCRIPTION:
Asthma affects 7 - 12 % of the population in North America and results in substantial morbidity and health care costs. Management of asthma is focused towards reducing airway inflammation through a combination of avoidance of inciting and triggering pro-inflammatory agents as well as anti-inflammatory medication. Corticosteroids and anti-leukotrienes are efficacious, but are neither universally effective nor free of side effects. Statins, which are currently widely prescribed and used safely to improve serum lipids and cholesterol, have anti-inflammatory properties which may be clinically useful in asthma either in addition to or perhaps instead of corticosteroids.

The objective of this research proposal is to conduct a randomized placebo controlled trial of 4 weeks statin therapy in patients in moderate to severe but stable asthma. We hypothesize that statins may directly reduce airway inflammation and/or contribute to the anti-inflammatory effects of corticosteroid treatment in these patients. We will measure the effects of statins by measuring airway sensitivity to methacholine, pulmonary function, sputum eosinophils, and quality of life in subjects with asthma after 4 weeks of treatment. Statins may become an alternative treatment option or act as steroid sparing agents in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Moderate to severe asthma based on Canadian Asthma Consensus Report
* Objective evidence of airway hyper-responsiveness (reversible airflow obstruction or positive methacholine challenge in previous two years
* On chronic maintenance inhaled corticosteroid therapy.

Exclusion Criteria:

* Asthma exacerbation within preceding 3 months necessitating any escalation of maintenance medications
* Chronic oral prednisone use
* Other respiratory, inflammatory and autoimmune disorder
* Abnormal baseline creatinine kinase, liver transaminases, or renal disease
* History of coronary artery disease, hyperlipidemia, or other condition requiring statin therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-02; Primary Completion 2013-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
PC20 Methacholine dose | 4 weeks

SECONDARY OUTCOMES:
Post bronchodilator FEV1 | 4 weeks
sputum eosinophil count | 4 weeks
daily dose of inhaled corticosteroid in beclomethasone disposable equivalents | 4 weeks
number of exacerbations or infections over the study period | 4 weeks
MiniAQLQ score (an asthma specific quality of life) | 4 weeks
liver enzymes | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diane Lougheed, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Background] Boulet LP, Becker A, Berube D, Beveridge R, Ernst P. Canadian Asthma Consensus Report, 1999. Canadian Asthma Consensus Group. CMAJ. 1999 Nov 30;161(11 Suppl):S1-61. PMID 10906907
- [Background] Weitz-Schmidt G. Statins as anti-inflammatory agents. Trends Pharmacol Sci. 2002 Oct;23(10):482-6. doi: 10.1016/s0165-6147(02)02077-1. PMID 12368073
- [Background] Pasternak RC, Smith SC Jr, Bairey-Merz CN, Grundy SM, Cleeman JI, Lenfant C; American College of Cardiology; American Heart Association; National Heart, Lung and Blood Institute. ACC/AHA/NHLBI Clinical Advisory on the Use and Safety of Statins. Circulation. 2002 Aug 20;106(8):1024-8. doi: 10.1161/01.cir.0000032466.44170.44. No abstract available. PMID 12186811